CLINICAL TRIAL: NCT00128544
Title: A Randomized, Blinded, Phase IIb Trial of Telbivudine (LdT) Versus the Combination of Telbivudine and Valtorcitabine (Val-LdC) in Patients With Chronic Hepatitis B
Brief Title: Telbivudine Versus the Combination of Telbivudine and Valtorcitabine in Patients With Chronic Hepatitis B
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Novartis (Industry)
Collaborators: Novartis Pharmaceuticals (Industry)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: NV-02C-004
Record Dates: First submitted 2005-08-08; First posted 2005-08-10 (Estimated); Last update posted 2017-06-16 (Actual); Status verified 2017-06

CONDITIONS: Hepatitis B
MeSH Terms: conditions — Hepatitis B | interventions — Telbivudine

INTERVENTIONS:
Drug: telbivudine
Drug: valtorcitabine

SUMMARY:
This study is being conducted to compare the effectiveness of the combination of valtorcitabine and telbivudine to telbivudine alone in patients with chronic hepatitis B.

ELIGIBILITY:
Inclusion Criteria:

* Clinical history compatible with compensated chronic hepatitis B

Other protocol-defined inclusion criteria may apply.

Exclusion Criteria:

* Patient is pregnant or breastfeeding
* Patient is co-infected with hepatitis C virus, hepatitis D virus or HIV
* Patient has previously received lamivudine, adefovir dipivoxil or an investigational anti-hepatitis B virus (HBV) nucleoside or nucleotide at anytime.

Other protocol-defined exclusion criteria may apply.

Ages: 18 Years to 70 Years | Sex: All
Age Groups: Adult, Older Adult
Enrollment: 130
Dates: Start 2005-05; Primary Completion 2007-05 (Actual); Study Completion 2007-05 (Actual)

CONTACTS AND LOCATIONS:
Locations (3):
- Pokfulam, Hong Kong
- Auckland, New Zealand
- Singapore, Singapore